CLINICAL TRIAL: NCT07185217
Title: Effects of Nurse Led Educational Intervention on Preventing Smart Phone Addiction Among Adolescent :A Health Belief Model Approach
Brief Title: Educational Intervention to Prevent Smartphone Addiction Among Adolescent
Acronym: smart phone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norther Private Collage of Nursing (Other)
Responsible Party: Principal Investigator, Amal Hashem, Associate professor, Norther Private Collage of Nursing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: smart phone addiction
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Smart Phone Addiction; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education intervention group (Active Comparator): the study group were divided into small groups 15-20 students. six session were needed for each group ,First session: it provide an overview of the educational intervention to enhance knowledge about smart phone addiction, Second session: it based on perceived susceptibility of the HBM , Third session: This session implemented based on the construct of perceived severity of HBM , Forth session: This session implemented based on the perceived benefits, perceived barriers, and perceived self-efficacy of the HBM. Fifth session: This session implemented based on cues to action, Session six: Three months after the fifth session, the post-intervention visit took place.
  Interventions: Other: class mate teaching subjects only
- control group (Sham Comparator): receive education classmate
  Interventions: Other: class mate teaching subjects only

INTERVENTIONS:
Other: class mate teaching subjects only — the participants receive educational classmate subjects.

SUMMARY:
The study aimed to evaluate the effect of nurse led educational intervention on preventing smart phone addiction among adolescent, participants were adolescents studying in prep school either in the first and second grades and their age ranged from 13- 16.

DETAILED DESCRIPTION:
The research hypothesis include adolescents who receive the nurse-led smartphone addiction prevention intervention based on health belief model in study group exhibit lower smartphone addiction level than those in control group.

-Adolescents who receive the nurse-led smartphone addiction prevention intervention based on health belief model had higher knowledge regarding smartphone addiction than those in control group.

Participants were divided into two groups (study and control). Both groups were asked to fill out all questionnaires before and after the study using the same tools. In the control group, adolescents receives routine care, and educational classes' only. Participants were asked to answer a post-test using the same pre-test questionnaires. And the study group were divided into small training groups with 15-20 participants and divided into small groups . Six sessions were needed for each group each session took about 1- 2hrs.

ELIGIBILITY:
Inclusion Criteria:

* their ages ranged between (13-16 years), and get acceptance from their parents to participate in the study.

Exclusion Criteria:

* students who unwilling to participates
* more than 16 years
* their parents refuse to participates

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
smartphone addiction level | eight month
  education intervention for prevention of smartphone addiction by using health belief model construct. by using smartphone addiction inventory , total score 104 mark, where high score indicate more smartphone addiction

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Egypt, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effectiveness of school-based interventions to reduce problematic digital technology use and screen time: A systematic review and meta-analysis — https://pmc.ncbi.nlm.nih.gov/articles/PMC12231446/